CLINICAL TRIAL: NCT00625898
Title: A Multicenter Phase III Randomized Trial of Adjuvant Therapy for Patients With HER2-Positive Node-Positive or High Risk Node-Negative Breast Cancer Comparing Chemotherapy Plus Trastuzumab With Chemotherapy Plus Trastuzumab Plus Bevacizumab
Brief Title: BETH Study: Treatment of HER2 Positive Breast Cancer With Chemotherapy Plus Trastuzumab vs Chemotherapy Plus Trastuzumab Plus Bevacizumab
Acronym: BETH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Cancer International Research Group (CIRG) (Other); Hoffmann-La Roche (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-44-I; CIRG (TRIO) 011 (Other: Cancer International Research Group); Roche BO20906 (Other: Roche); BETH (Other: NSABP)
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: HER2 positive breast cancer; invasive breast cancer; bevacizumab; NSABP; Roche; CIRG; trastuzumab; cyclophosphamide; docetaxel; carboplatin; 5-fluorouracil; epirubicin
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Trastuzumab; Carboplatin; Bevacizumab; Fluorouracil; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1A: TCH-H (Active Comparator): Docetaxel (T), Carboplatin (C), and Trastuzumab (H) followed by Trastuzumab (H)
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: Carboplatin
- 1B: TCHB-HB (Experimental): Docetaxel (T), Carboplatin (C), Trastuzumab (H), Bevacizumab (B) followed by Trastuzumab (T) and Bevacizumab (B)
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: Carboplatin; Drug: Bevacizumab
- 2A: TH-FEC-H (Active Comparator): Docetaxel (T) and Trastuzumab (H) followed by 5-fluorouracil (F), Epirubicin (E), and Cyclophosphamide (C) followed by Trastuzumab (H)
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide
- 2B: THB-FEC-HB (Experimental): Docetaxel (T), Trastuzumab (H), and Bevacizumab (B) followed by 5-Fluorouracil (F), Epirubicin (E), and Cyclophosphamide (C) followed by Trastuzumab (H) and Bevacizumab (B)
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: Bevacizumab; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 IV on day 1 every 3 weeks for cycles 1-6, Arms 1A and 1B
  100 mg/m2 on day 1 every 3 weeks for cycles 1-3, Arms 2A and 2B
  Other Names: Taxotere
Drug: Trastuzumab — First dose: 8 mg/kg IV on day 1 of cycle 1 only. Subsequent doses: 6 mg/kg IV on day 1 every 3 weeks for cycles 2-6. Following completion of chemotherapy cycles: 6 mg/kg IV every 3 weeks until 1 year following first trastuzumab dose. Arms 1A and 1B
  First dose: 8 mg/kg IV on day 1 of cycle 1 only. Subsequent doses: 6 mg/kg IV on day 1 every 3 weeks for cycles 2-3. 21 days after last dose of FEC: 8 mg/kg IV first post-FEC dose only; subsequent doses 6 mg/kg IV every 3 weeks for a total of 1 year. Arms 2A and 2B
  Other Names: Herceptin
Drug: Carboplatin — 6 mg/ml/min IV on day 1 every 3 weeks for cycles 1-6
  Arms: 1A: TCH-H; 1B: TCHB-HB
Drug: Bevacizumab — 15 mg/kg IV on day 1 every 3 weeks for cycles 1-6. Following completion of chemotherapy cycles: 15 mg/kg IV on day 1 every 3 weeks until 1 year following first bevacizumab dose. Arm 1B
  15 mg/kg IV on day 1 every 3 weeks for cycles 1-3. 21 days after the last dose of FEC: 15 mg/kg IV on day 1 every 3 weeks until 1 year following first bevacizumab dose. Arm 2B
  Other Names: Avastin
  Arms: 1B: TCHB-HB; 2B: THB-FEC-HB
Drug: 5-Fluorouracil — 600 mg/m2 IV on day 1 every 3 weeks for cycles 4-6
  Arms: 2A: TH-FEC-H; 2B: THB-FEC-HB
Drug: Epirubicin — 90 mg/m2 IV on day 1 every 3 weeks for cycles 4-6
  Arms: 2A: TH-FEC-H; 2B: THB-FEC-HB
Drug: Cyclophosphamide — 600 mg/m2 IV on day 1 every 3 weeks for cycles 4-6
  Arms: 2A: TH-FEC-H; 2B: THB-FEC-HB

SUMMARY:
The trial will determine the value of adding bevacizumab to chemotherapy plus trastuzumab in patients with resected node-positive or high risk node-negative, HER2-positive breast cancer.

DETAILED DESCRIPTION:
This Phase III, randomized, open-label trial will determine whether the regimens of chemotherapy plus trastuzumab plus bevacizumab improve invasive disease-free survival (IDFS) relative to the regimens of chemotherapy plus trastuzumab. Secondary aims include determining whether the addition of bevacizumab to chemotherapy plus trastuzumab will improve disease-free survival (DFS), overall survival (OS), recurrence-free interval (RFI), and distant recurrence-free interval (DRFI). The benefit of adding bevacizumab for IDFS, DFS, OS, RFI, and DRFI will also be evaluated for each of the two chemotherapy regimens. The cardiac and non-cardiac toxicities of each of the regimens will also be evaluated.

Following local determination that the tumor is HER2-positive for gene amplification by in situ hybridization or is IHC 2+ or 3+, a tumor sample must be submitted for HER2 testing by a designated central laboratory. If central testing confirms that the tumor is HER2-positive (either positive by FISH or IHC 3+) and all other eligibility criteria have been met, the patient will be randomized to a regimen of chemotherapy and trastuzumab with or without bevacizumab.

Patients in the trial will be enrolled in one of two chemotherapy regimen cohorts. One cohort will receive 6 cycles of docetaxel/carboplatin plus trastuzumab (TCH) with or without bevacizumab; the other cohort will receive 3 cycles of docetaxel plus trastuzumab given with or without bevacizumab followed by 3 cycles of 5-Fluorouracil, Epirubicin, Cyclophosphamide (TH-FEC). With both regimens, patients will continue trastuzumab with or without bevacizumab following chemotherapy to complete 1 year of targeted therapy. Following completion of chemotherapy, patients will also receive adjuvant radiotherapy and endocrine therapy as clinically indicated.

The trial will be conducted by investigators affiliated with the Cancer International Research Group (CIRG) and the National Surgical Adjuvant Breast and Bowel Project (NSABP). CIRG and NSABP investigators will only enroll patients in the TCH regimen cohort. Additional investigators, referred to in the protocol as Independent Investigators, will enroll patients in both the TCH regimen or the TH-FEC regimen cohort depending on institutional preference for the one regimen that will be used by that institution for the duration of the trial.

Patients will be given the option of allowing their tumor samples to be used for the BETH translational research and correlative science studies. Also, patients will be asked to consent to the submission of blood and serum samples at scheduled time points during the study.

LVEF assessments will be performed before study entry and then at scheduled time points during therapy and at 18, 36, and 60 months following randomization.

The planned sample size for the trial is 3,000 patients randomized in the faster accruing cohort and a minimum of 3,500 patients overall.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 10 years, excluding their diagnosis of breast cancer.
* Women who have had breast reconstruction utilizing tissue expanders must be in agreement with delaying surgery to replace the tissue expanders with permanent implants until 3 months following the last dose of bevacizumab
* Women of reproductive potential must agree to use an effective non-hormonal method of contraception (for example condoms, some intrauterine devices, diaphragms, vasectomized partner, or abstinence) during therapy and for at least 6 months after the last dose of bevacizumab and/or trastuzumab.
* Submission of tumor samples from the breast surgery for central HER2 testing is required for all patients prior to enrollment in the BETH Trial
* Signed and dated IRB/EC-approved consent
* ECOG performance status of 0 or 1
* The tumor must be unilateral invasive adenocarcinoma of the breast on histologic examination.
* The breast cancer must be HER2-positive based on test results as follows: Local testing (if available) should demonstrate that the tumor is IHC 2+ or 3+ or is considered to be HER2-positive for gene amplification by FISH, CISH, or other in situ hybridization (ISH) method. If local ISH test results are considered equivocal, the tumor can be submitted for central HER2 testing. (If local testing is not possible, the tumor can be submitted for central HER2 testing.) Central testing (a requirement for ALL patients) must demonstrate that the tumor is HER2-positive which is defined as FISH-positive and/or IHC 3+.
* All of the following staging criteria (according to the 6th edition of the AJCC Cancer Staging Manual) must be met: By pathologic evaluation, primary tumor must be pT1-3; By pathologic evaluation, ipsilateral nodes must be pN0, pN1 (pN1mi, pN1a, pN1b, pN1c), pN2a, pN3a, or pN3b. If pN0, at least one of the following criteria must be met: Pathologic tumor size > 2.0 cm; ER negative and PgR negative; Histologic and/or nuclear grade 2 (intermediate) or 3 (high); or Age < 35 years
* Patients must have undergone either a total mastectomy or breast conserving surgery (lumpectomy).
* For patients who undergo lumpectomy, the margins of the resected specimen must be histologically free of invasive tumor and ductal carcinoma in situ (DCIS) as determined by the local pathologist. If pathologic examination demonstrates tumor at the line of resection, additional operative procedures may be performed to obtain clear margins. If tumor is still present at the resected margin after re-excision(s), the patient must undergo total mastectomy to be eligible. (Patients with margins positive for lobular carcinoma in situ [LCIS] are eligible without additional resection.)
* For patients who undergo mastectomy, margins must be free of gross residual tumor. Patients with microscopic positive margins are eligible.
* Patients must have completed one of the following procedures for evaluation of pathologic nodal status: Sentinel lymphadenectomy followed by removal of additional non-sentinel lymph nodes if the sentinel node (SN) is positive; Sentinel lymphadenectomy alone if pathologic nodal staging based on sentinel lymphadenectomy is pN0, pN1mi or pN1b; or Axillary lymphadenectomy without SN isolation procedure.
* The interval between the last surgery for breast cancer (treatment or staging) and randomization must be at least 28 days but no more than 84 days.
* Patients must have ER analysis performed on the primary tumor prior to randomization. If ER analysis is negative, then PgR analysis must also be performed.
* The most recent postoperative blood counts, performed within 6 weeks prior to randomization, must meet the following criteria: ANC must be greater than or equal to 1200/mm3; Platelet count must be greater than or equal to 100,000/mm3; and Hemoglobin must be greater than or equal to 10 g/dL.
* The following criteria for evidence of adequate hepatic function must be met based on the results of the most recent postoperative tests performed within 6 weeks prior to randomization: total bilirubin must be less than or equal to upper limit of normal (ULN) for the lab unless the patient has a bilirubin elevation > ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and alkaline phosphatase must be less than or equal to 2.5 x ULN for the lab; and AST must be less than or equal to 1.5 x ULN for the lab. Alkaline phosphatase and AST may not both be > the ULN.
* Patients with AST or alkaline phosphatase > ULN are eligible for inclusion in the study if liver imaging (CT, MRI, PET scan, or PET-CT scan performed within 3 months prior to randomization) does not demonstrate metastatic disease and the requirements for evidence of adequate hepatic function are met.
* Patients with alkaline phosphatase that is > ULN but less than or equal to 2.5 x ULN are eligible for inclusion in the study if a bone scan,PET scan, or PET-CT scan (performed within 3 months prior to randomization) does not demonstrate metastatic disease.
* The following criteria for renal function must be met based on the results of the most recent postoperative tests performed within 6 weeks prior to randomization: Serum creatinine must be less than or equal to ULN for the lab. Measured or calculated creatinine clearance must be > 60 mL/min.
* A urine sample must be tested for protein by determination of the urine protein/creatinine (UPC) ratio or by urine dipstick. UPC ratio must be less than 1.0. Urine dipstick must indicate 0-1+ protein. If dipstick reading is greater than or equal to 2+, determine the UPC ratio, which must be less than 1.0, or collect a 24-hour urine specimen, which must demonstrate < 1.0 g of protein per 24 hours.
* LVEF assessment must be performed within 3 months prior to randomization. The LVEF must be greater than or equal to 55% regardless of the cardiac imaging facility's lower limit of normal (LLN).
* The ECG (performed within 3 months prior to randomization) must not have demonstrated any of the following conditions: ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; and conduction abnormality requiring a pacemaker.

Exclusion Criteria:

* Inflammatory breast cancer.
* Definitive clinical or radiologic evidence of metastatic disease. (Chest imaging [mandatory for all patients] and other imaging [if required] must have been performed within 3 months prior to randomization.)
* Synchronous or previous contralateral invasive breast cancer (Patients with synchronous or previous contralateral DCIS or LCIS are eligible).
* History of ipsilateral invasive breast cancer regardless of treatment or ipsilateral DCIS treated with excision and RT. (Patients with history of ipsilateral LCIS are eligible.)
* History of non-breast malignancies within the 5 years prior to study entry, except for the following: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinomas of the skin.
* Previous therapy with anthracyclines, taxanes, carboplatin, trastuzumab, or bevacizumab for any malignancy.
* RT, chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to randomization.
* Continued therapy with any hormonal agent such as raloxifene or tamoxifen (or other SERM) or an aromatase inhibitor. (Patients are eligible if these medications are discontinued prior to randomization.)
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy, etc. Patients are eligible if these medications are discontinued prior to randomization.
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens. This includes but is not confined to: Active cardiac disease - angina pectoris that requires the use of anti-anginal medication; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromise in cardiac function; and symptomatic pericarditis. History of cardiac disease - myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LV function; history of documented CHF; and documented cardiomyopathy.
* Uncontrolled hypertension defined as systolic blood pressure (BP) > 150 mmHg or diastolic BP > 90 mmHg, with or without anti-hypertensive medication. (BP must be assessed within 28 days prior to randomization.) Patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria.
* History of hypertensive crisis or hypertensive encephalopathy.
* History of TIA or CVA.
* History of any arterial thrombotic event within 12 months before randomization.
* Symptomatic peripheral vascular disease.
* Intrinsic lung disease resulting in dyspnea.
* Unstable diabetes mellitus.
* Active infection or chronic infection requiring chronic suppressive antibiotics.
* Any significant bleeding within 6 months before randomization, exclusive of menorrhagia in premenopausal women.
* Non-healing wound, skin ulcers, or incompletely healed bone fracture.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to planned start of study therapy.
* Anticipation of need for major surgical procedures during study therapy and for at least 3 months following completion of bevacizumab.
* Gastroduodenal ulcer(s) documented by endoscopy to be active within 6 months before randomization.
* History of GI perforation, abdominal fistulae, or intra-abdominal abscess.
* Known bleeding diathesis or coagulopathy.
* Requirement for therapeutic doses of coumadin or equivalent.
* Sensory/motor neuropathy greater than or equal to grade 2, as defined by the NCI CTCAE v3.0.
* Conditions that would prohibit administration of corticosteroids.
* Chronic daily treatment with corticosteroids (dose of > 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids).
* History of hypersensitivity reaction to drugs formulated with polysorbate 80.
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing must be performed within 14 days prior to randomization according to institutional standards for women of child-bearing potential.)
* Other non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Use of any investigational product within 4 weeks prior to enrollment in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3509 (Actual)
Dates: Start 2008-04; Primary Completion 2013-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (IDFS) | up to 10 years

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) within chemotherapy cohorts | up to 10 years
Disease-free survival (DFS) | up to 10 years
Overall survival (OS) | Time from randomization until death from any cause or up to a maximum of 10 years from study entry
Recurrence-free interval (RFI) | Time from randomization until local, regional or distant recurrence or up to a maximum of 10 years from study entry
Distant recurrence-free interval (DRFI) | Time from randomization until distant disease recurrence only or up to a maximum of 10 years from study entry
Cardiac toxicity. Cumulative incidence of severe cardiac events defined as definite or probable cardiac death, or NYHA Class III or IV CHF | 2-3 weeks after cycle 3; 2-3 weeks after last chemotherapy dose; 7, 10, 18, 36, and 60 months from randomization
Non-cardiac toxicity. Frequencies of adverse events categorized using the NCI CTCAE v3.0. | within 3 days of each chemotherapy cycle; 2-3 weeks following last chemotherapy dose; every 6 weeks during targeted therapy; every 6 months through year 5; every 12 months years 6 - 10
Identification of biomarkers (from tumor and serum/plasma) predictive for the level of benefit from the addition of bevacizumab to standard adjuvant systemic treatment for HER2-positive breast cancer as well as for cardiac toxicity | baseline, during therapy and follow-up, within 2 weeks of LVEF assessments, any protocol-specified cardiac event, and after diagnosis of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (647):
- United States (391):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Clearview Cancer Institute-Decatur, Decatur, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Clearview Cancer Institute- Huntsville, Huntsville, Alabama
  - Northern Arizona Hematology & Onclogy Associates, Flagstaff, Arizona
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Central Hematology/Oncology Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - Hematology-Encinitas, Encinitas, California
  - Scripps Clinic Encinitas, Encinitas, California
  - Kaiser Permanente-Fontana, Fontana, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Breastlink Medical Group, Inc, Hawthorne, California
  - Pacific Shores Medical Group, Huntington Beach, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Hematology-La Jolla, La Jolla, California
  - Sabina R. Wallach, MD., AMC, La Jolla, California
  - Scripps Cancer Center-San Diego, La Jolla, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Kaiser Permanente-Sunset, Los Angeles, California
  - Kaiser Permanente-West Los Angeles, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - North County Oncology Medical Clinic, Inc., Oceanside, California
  - Kaiser Permanente-Panorama City, Panorama City, California
  - Kaiser Permanente-Orange County, Panorama City, California
  - Wilshire Oncology Medical Group, Pasadena, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente-Sacramento, Roseville, California
  - Sutter Medical Center, Sacramento, California
  - Sutter Medical Group, Sacramento, California
  - Peter T. Reissman, MD, Inc, San Diego, California
  - William Stanton, MD, Inc, San Diego, California
  - Kaiser Permanente-San Diego, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Scripps Clinic-Rancho Bernardo, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Hayward, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Santa Barbara, California
  - Kaiser Permanente-Santa Clara, Santa Clara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - UCLA/Santa Clarita Valley Cancer Center, Valencia, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - San Diego Pacific Oncology & Hematology-Vista, Vista, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Cypress Hematology/Oncology, Denver, Colorado
  - Rocky Mountain Cancer Center - Midtown, Denver, Colorado
  - CCOP-Colorado Cancer Research Prog. Inc.(Administrative Only), Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente Rock Creek, Lafayette, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Oncology Associates P.C.-Avon, Avon, Connecticut
  - Medical Specialists of SWIM, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Medical Specialists of Fairfield, Fairfield, Connecticut
  - Oncology Associates of Bridgeport-Fairfield, Fairfield, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Connecticut Multi Specialty Group-Hartford, Hartford, Connecticut
  - Oncology Associates P.C.-Hartford, Hartford, Connecticut
  - Medical Oncology and Hematology, P.C., Meriden, Connecticut
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Black Rock Medical Group, Trumbull, Connecticut
  - Oncology Associates of Bridgeport-Trumbull, Trumbull, Connecticut
  - Medical Oncology & Hematology, P.C., Waterbury, Connecticut
  - Connecticut Multi Specialty Group-Wethersfield, Wethersfield, Connecticut
  - Oncology Associates P.C.-Willimantic, Willimantic, Connecticut
  - CCOP, Christiana Care Health Services Inc., Newark, Delaware
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Washington Oncology-Hematology Center, PC-Washington, Washington D.C., District of Columbia
  - Lynn Cancer Institute, Boca Raton, Florida
  - Florida Cancer Specialists-Bonita Springs, Bonita Springs, Florida
  - Florida Cancer Specialists-Bradenton, Bradenton, Florida
  - Florida Cancer Specialists, Brandon, Brandon, Florida
  - Florida Cancer Specialists-Cape Coral Parkway, Cape Coral, Florida
  - Florida Cancer Specialists-Cape Coral Del Prado, Cape Coral, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists-Englewood, Englewood, Florida
  - Florida Cancer Specialists-Fort Myers Broadway, Fort Myers, Florida
  - Florida Cancer Specialists-Fort Myers Summerlin, Fort Myers, Florida
  - Robert R. Carroll, MD, PA, Gainesville, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Florida Cancer Specialists-Naples Goodlette, Naples, Florida
  - Florida Cancer Specialists-NAPA Ridge, Naples, Florida
  - Integrated Community Oncology Network, Orange Park, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists, Cornerstone, Palm Harbor, Florida
  - Florida Cancer Specialists-Port Charlotte, Port Charlotte, Florida
  - Florida Cancer Specialist-Cattleman, Sarasota, Florida
  - Florida Cancer Specialists-Downtown, Sarasota, Florida
  - Florida Cancer Specialists-Park Place, St. Petersburg, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists-Venice Island, Venice, Florida
  - Florida Cancer Specialists-Venice, Venice, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Grady Healthsystem, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Augusta Oncology Associates, Augusta, Georgia
  - Northwest Georgia Oncology Centers PC, Austell, Georgia
  - Northwest Georgia Oncology Centers PC, Carrollton, Georgia
  - Northwest Georgia Oncology Centers PC, Cartersville, Georgia
  - Suburban Hematology-Oncology Associates, Lawrenceville, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Georgia Cancer Specialists, Macon, Georgia
  - Georgia Cancer Specialists, Marietta, Georgia
  - Suburban Hematology Oncology Associates PC, Snellville, Georgia
  - Oncare Hawaii, Inc-POB2, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Oncare Hawaii, Inc-KMP, Honolulu, Hawaii
  - Kootenai Cancer Center, Coeur d'Alene, Idaho
  - Mountain States Tumor Institute, Meridian, Idaho
  - Mountain States Tumor Institute, Twin Falls, Idaho
  - Cancer Care & Hematology Specialists of Chicagoland, Arlington, Illinois
  - MBCCOP, John H. Stroger, JR., Hospital of Cook County-Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Crossroads Cancer Center, Decatur, Illinois
  - Cancer Care Specialists-Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Edward Hospital, Naperville, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland, Winfield, Illinois
  - Yorkville Family Practice, Yorkville, Illinois
  - Cancer Care of Southern Indiana, Bloomington, Indiana
  - Corydon Hospital Medical Plaza, Corydon, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology-Oncology, P.C. (Elkhart), Elkhart, Indiana
  - Waverly Hematology Oncology, Gary, Indiana
  - Clark Medical Building, Jeffersonville, Indiana
  - Howard Regional Health System, Kokomo, Indiana
  - Michiana Hematology-Oncology, P.C. (LaPorte), La Porte, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Michiana Hematology-Oncology PC, Plymouth, Indiana
  - Oncology, P.C. Plymouth, Plymouth, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology-Oncology, P.C. (Main Office), South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology-Oncology, P.C. Cedar St., South Bend, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Hematology and Medical Oncology Consultants-Bettendorf, Bettendorf, Iowa
  - Hematology and Medical Oncology Consultants-Davenport, Davenport, Iowa
  - University of Iowa, Iowa City, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - NortonHealthcare Pavillion, Louisville, Kentucky
  - Norton Medical Plaza II, Louisville, Kentucky
  - Norton Medical Plaza West, Louisville, Kentucky
  - Old Brownsboro Crossing, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Harry & Jeannette Weinberg Cancer Institute, Baltimore, Maryland
  - Hematology-Oncology Associates, Baltimore, Maryland
  - Carolyn Hendricks, MD, Bethesda, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - The Office of Frederik Smith, Chevy Chase, Maryland
  - Washington Oncology-Hematology Center, PC-Chevy Chase, Chevy Chase, Maryland
  - Associates in Oncology/Hematology, Rockville, Maryland
  - Peninsula Regional Oncology & Hematology, Salisbury, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Oncology Care Associates, Wheaton, Maryland
  - Berkshire Hematology Oncology, P.C.-North Adams, North Adams, Massachusetts
  - Berkshire Hematology Oncology, P.C., Pittsfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - CCOP, St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Battle Creek Health System, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Dr. Cook and Abramson - Bay City, Bay City, Michigan
  - St. Joseph Mercy Woodland Health Center, Brighton, Michigan
  - Josephone Ford Cancer Center, Brownstown, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - UP Hematology/Oncology Assoc.-Doctor's Park Family Physicians, Escanaba, Michigan
  - CCOP Hurley Medical Center, Flint, Michigan
  - Genesys Hurley, Flint, Michigan
  - Sing and Arora, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - St. Mary's Health Services, Grand Rapids, Michigan
  - CCOP, St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Portage Internal Medical Associates, Hancock, Michigan
  - UP Hematology/Oncology Associates, Iron Mountain, Michigan
  - UP Hematology/Oncology Associates-Gogebic Range, Ironwood, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Hematology/Oncology Associates of OH and MI, PC, Lambertville, Michigan
  - CCOP, Sparrow Health System, Lansing, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - Hematology Oncology-Lapeer, Lapeer, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - Keewanaw Memorial Hospital, Laurium, Michigan
  - St. Mary Mercy Hospital - Livonia, Livonia, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Upper Peninsula Hematology/Oncology Associates, Marquette, Michigan
  - Community Cancer Care Specialists-Mt. Clemens, Mount Clemens, Michigan
  - Mount Clemens Regional Medical Center, Mount Clemens, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Michiana Hematology-Oncology PC, Niles, Michigan
  - CCOP, William Beaumont Hospital, Royal Oak, Michigan
  - CCOP, St. Mary's Medical Center, Saginaw, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Michiana Hematology-Oncology, PC Lakeland, Saint Joseph, Michigan
  - Chippewa Medical Associates, Sault Ste. Marie, Michigan
  - Osteopathic Medical Oncology Hematology, Shelby, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - CCOP, St. John Macomb Hospital, Warren, Michigan
  - Henry Ford Medical Center-West Bloomfield, West Bloomfield, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Minnesota Oncology Hematology-Burnsville, Burnsville, Minnesota
  - Park Nicollet Clinic, Burnsville, Minnesota
  - Hubert H. Humphrey Cancer Center - Coon Rapids, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology-Edina, Edina, Minnesota
  - Fairview Southdale Medical Oncology Clinic, Edina, Minnesota
  - Hubert H. Humphrey Cancer Center - Fridley, Fridley, Minnesota
  - Minnesota Oncology Hematology PA - Maplewood, Maplewood, Minnesota
  - Minnesota Oncology Hematology-Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center-Robbinsdale, Robbinsdale, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Minnesota Hematology Oncology-St. Paul, Saint Paul, Minnesota
  - Minnesota Oncology Hematology-Waconia, Waconia, Minnesota
  - Minnesota Oncology Hematology, Woodbury, Minnesota
  - University of Tennessee Cancer Institute, Southaven, Mississippi
  - University of Missouri-Ellis Fischel, Columbia, Missouri
  - Freeman Cancer Institute, Joplin, Missouri
  - St. John's Regional Health Center-Joplin, Joplin, Missouri
  - Saint Luke's Hospital, Kansas City, Missouri
  - CCOP, Kansas City (Administrative Only), Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Cox Health Systems, Springfield, Missouri
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Comprehensive Cancer Centers of Nevada (Siena), Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists- Shadow Lane, Las Vegas, Nevada
  - Cancer Consultants, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Alpine Hematology-Oncology, Reno, Nevada
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Drs. Forte, Schleider, Attas and Condemi, PA, Englewood, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - New York Oncology Hematology PC-Albany, Albany, New York
  - NY Oncology Hematology PC at Albany Medical Center, Albany, New York
  - Amsterdam Community Cancer Program, Amsterdam, New York
  - Interlakes Oncology & Hematology, P.C., Canandaigua, New York
  - Hematology Oncology Assaociates of CNY, CCOP, East Syracuse, New York
  - NY Oncology Hematology PC-Hudson Carvell Cancer Tx Prog., Hudson, New York
  - NY Oncology Hematology PC- Latham- Capital District Oncology Hematology, Latham, New York
  - Beth Israel Medical Center, New York, New York
  - St. Luke's-Roosevelt Hospital Center, New York, New York
  - Riverview Cancer Care Medical Association, Rexford, New York
  - Hematology Oncology Associates of CNY, CCOP, Rome, New York
  - University Hospital and Medical Center - SUNY, Stony Brook, New York
  - University Hospital and Medical Center-SUNY, Stony Brook, New York
  - Hematology Oncology Assoc. of CNY, CCOP (Comm. General Hospital Satellite Office), Syracuse, New York
  - Troy Cancer Treatment Program, Troy, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - CCOP, Mission Hospitals, Inc., Asheville, North Carolina
  - Cancer Center of NC at Asheville, Asheville, North Carolina
  - Carolinas Hematology-Oncology Associates - Tyron St, Charlotte, North Carolina
  - Carolinas Medical Center - Blumenthal Cancer Center, Charlotte, North Carolina
  - CCOP Presbyterian Hospital, Charlotte, North Carolina
  - Mecklenburg Medical Group - Morehead Medical Dr, Charlotte, North Carolina
  - Mecklenburg Medical Group - Cameron Valley Pkwy, Charlotte, North Carolina
  - Carolinas Hematology Oncology Associates - Harris Blvd., Charlotte, North Carolina
  - Carolinas Hematology-Oncology - John J. Delaney, Charlotte, North Carolina
  - CCOP, Wayne Memorial Hospital, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center, Greensboro, North Carolina
  - Northwestern Carolina Oncology & Hematology, PA, Hickory, North Carolina
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Alliance Cancer Center, Alliance, Ohio
  - Aultman Hospital, Canton, Ohio
  - Tri County Hematology/Oncology, Canton, Ohio
  - Kenwood Office, Cincinnati, Ohio
  - Oncology/Hematology Care Clinical Trials LLC, Cincinnati, Ohio
  - North Treatment Center - Blue Ash Medical Center, Cincinnati, Ohio
  - Oncology/Hematology Care Clinical Trials LLC, Cincinnati, OH Blue Ash Med. Cntr. (Administrative Only), Cincinnati, Ohio
  - Case Western Reserve/University Hospitals-Ireland Cancer Cntr., Cleveland, Ohio
  - Dayton Physicians-LLC-Hematology & Medical Oncology Division, Dayton, Ohio
  - Healthplex, Fairfield, Ohio
  - Dayton Physicians, LLC - Greenville, Greenville, Ohio
  - Hamilton Office, Hamilton, Ohio
  - Dayton Clinical Oncology Program-Kettering, Kettering, Ohio
  - Marian A. Llenado Lee, MD, Inc., Kettering, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - UHHS - Chagrin Highlands, Orange, Ohio
  - UHHS Green Road-Ireland Cancer Center, South Euclid, Ohio
  - Flower Memorial Hospital, Sylvania, Ohio
  - Bayview Oncology Associates, Toledo, Ohio
  - Toledo Clinic, Toledo, Ohio
  - UHHS Westlake-Ireland Cancer Center, Westlake, Ohio
  - Northwest Cancer Specialists-Portland, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Northwest Cancer Specialists-Adventist Office, Portland, Oregon
  - CCOP, Columbia River Oncology, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - Hematology Oncology Associates of NE PA, Donora, Pennsylvania
  - Ephrata Cancer Center at Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Cancer Centers Arnold Palmer Pavilion-Mountainview, Greensburg, Pennsylvania
  - UPMC Cancer Centers Arnold Palmer-Oakbrook, Greensburg, Pennsylvania
  - UPMC Cancer Centers-Indiana, Indiana, Pennsylvania
  - UPMC Cancer Centers-John P. Murtha Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Centers - McKeesport Hospital, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Cancer Centers Arnold Palmer-Mt. Pleasant, Mount Pleasant, Pennsylvania
  - Kimmel Cancer Center at Jefferson, Philadelphia, Pennsylvania
  - Cancer Center at Center One, Philadelphia, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Allegheny General Hospital/Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - NSABP Foundation, Inc, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers - UPMC Passavant, Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Hematology and Oncology Associates, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - UPMC Cancer Centers-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Centers - Wexford, Wexford, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Thompson Oncology Group-Blount, Knoxville, Tennessee
  - Thompson Cancer Survival Center-Dowell Springs, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Oncology Group-West, Knoxville, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Texas Oncology- Sammons CC, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Covenant Health System dba Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center, St. George, Utah
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - MBCCOP, Virginia Commonwealth University, Richmond, Virginia
  - Overlake Internal Medicine, Bellevue, Washington
  - Rockwood Cancer Treatment Center - Sinto Ave, Spokane, Washington
  - Rockwood Cancer Treatment Center, Spokane, Washington
  - Southwest Washington Hospital, Vancouver, Washington
  - Northwest Cancer Specialists-136th Ave, Vancouver, Washington
  - Northwest Cancer Specialists-134th St., Vancouver, Washington
  - West Virginia University Hospitals Inc., Morgantown, West Virginia
  - Oncology Alliance-Burlington, Burlington, Wisconsin
  - Oncology Alliance-Franklin, Franklin, Wisconsin
  - Oncology Alliance, Glendale, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Oncology Alliance-Kenosha South, Kenosha, Wisconsin
  - Oncology Alliance-Kenosha North, Kenosha, Wisconsin
  - CCOP, Marshfield Clinic, Marshfield, Wisconsin
  - Oncology Alliance-Menomonee Falls, Menomonee Falls, Wisconsin
  - Oncology Alliance-Mequon, Mequon, Wisconsin
  - Oncology Alliance-South, Milwaukee, Wisconsin
  - Oncology Alliance-Racine, Racine, Wisconsin
  - Oncology Alliance-Waukeska, Waukesha, Wisconsin
  - Marshfield Clinic Weston Center, Weston, Wisconsin
- Argentina (5):
  - Breast Clinica de la mama, La Plata, Buenos Aires
  - Hospital Universitario Austral, Presidente Derqui, Buenos Aires
  - Centro Oncologico Rosario (COR), Rosario, Sante Fe
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - CEMIC, Buenos Aires
- Australia (14):
  - Macarthur Cancer Center, Campbelltown, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Cancer Therapy Center, Liverpool, New South Wales
  - North Shore Private Hospital, St Leonards, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Southern Medical Day Care, Wollongong, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Ashford Cancer Center, Ashford, South Australia
  - Flinders Medical Centre, Bedford, South Australia
  - Frankston Hospital, Frankston, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Mount Medical Center, Perth, Western Australia
  - Berdat Family Comprehensive Cancer Centre, Subiaco, Western Australia
- Austria (13):
  - Krankenhaus Barmherzige Brueder Graz, Medizinische Abteilung, Graz
  - Universitatsfrauenklinik Graz, Graz
  - Medizinische Universitat Graz - Onkologie, Graz
  - AI University Hospital Innsbruck, Innsbruck
  - Bezirkskrankenhaus Kufstein, Innere Medizin, Kufstein
  - Landeskrankenhaus Leoben, Abteilung fur Haemato-Onkologie, Leoben
  - Krankenhaus Barmherzige Schwestern Linz, Kooperative Studiengruppe, Chirurgie, Linz
  - AI Universitätsklinikum der PMU Landeskliniken, Salzburg
  - AKH Vienna, Vienna
  - Medizinische Universitaet Wien-Allgemeines Krankenhaus, Onkologie, Vienna
  - Krankenhaus Hietzing, Gynaekologische Abteilung, Vienna
  - Landeskrankenhaus Voecklabruck, 2. Medizinische Abteilung, Vöcklabruck
  - Klinikum Wels-Grieskirchen, Kooperative Gruppe Wels/4. Medizinische Abteilung, Wels
- Belgium (4):
  - AZ Klina, Brasschaat
  - C. H. Notre-Dame and Reine Fabiola, Charleroi
  - Clinique St Pierre, Ottignies
  - Medical Institute St. Augustinus, Wilrijk
- Clinical Centre University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- Brazil (13):
  - Centro Goiano de oncologia, Goiânia, Goiás
  - Lifecenter Sistema de Saude S/A, Belo Horizonte, Minas Gerais
  - Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro
  - Clinica Oncologistas Associados, Rio de Janeiro, Rio de Janeiro
  - Assoiacao hospital de caridade de ijui, Ijuí, Rio Grande do Sul
  - Hospital Das Clinicas de Porto Alegre-HCPA, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericoria de Porto Alegre Nucleo de Novos Tratamentos, Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundacao Dr. Amaral Carvalho, Jaú, São Paulo
  - Instituto de Oncologia Clinica de Piracicaba, Piracicaba, São Paulo
  - Centro de Oncologia e Hematologia da Faculdade de Medicina do ABC, Santo André, São Paulo
  - Instituto do Cancer de Sao Paulo, São Paulo, São Paulo
  - Conjunto Hospitalar de Sorocaba, Sorocaba
- Bulgaria (2):
  - District Oncology Dispensary Plovdiv, Plovdiv
  - MHAT "Tsaritsa Yoanna-ISUL" EOOD, Sofia
- Canada (19):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Dept of Medicine, Edmonton, Alberta
  - Lion's Gate Hospital, North Vancouver, British Columbia
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - William Osler Health Center, Brampton, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - St. Michaels Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hospital du Sacre-Coeur, Montreal, Quebec
  - University of Montreal Hospital Group, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire De Quebec, Hospital du St-Sacrement, Québec, Quebec
- Hospital Regional Rancagua, Rancagua, Región del Libertador General Bernardo O’Higgins, Chile
- China (10):
  - Chinese Academy of Medical Science, Beijing
  - The Pla 307 Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Fuzhou General Hospital of Nanjing Military Area, Fuzhou
  - Sun Yat-sen University Hospital, Guangzhou
  - 1st Affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Tumor Hospital, Hangzhou
  - Tianjin Cancer Hospital, Tianjin
- University Hospital Zagreb, Zagreb, Croatia
- FN Na Bulovce, Prague, Czechia
- National Cancer Institute, Cairo, Egypt
- Tartu University Hospital Clinic of Hematology and Oncology, Tartu, Estonia
- France (22):
  - CHU D'Amiens, Amiens
  - CH-Service Hemato-Oncologie, Beauvais
  - Clinique Bordeaux Nord Aquitaine, Bordeaux
  - CHU Morvan, Brest
  - Hopital Pasteur, Colmar
  - Ch intercommunal de creteil, Créteil
  - Centre Leonard de Vinci, Dechy
  - Institut Daniel Hollard, Grenoble
  - CHD les Oudairies, La Roche-sur-Yon
  - Clinique Francois Chenieux, Limoges
  - CHU Dupuytren, Limoges
  - Hopital St. Joseph, Marseille
  - Centre Regional de Lutte contre le Cancer (CRLC) Val d'Aurelle, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Clinique Hartmann, Neuilly-sur-Seine
  - CHU Hotel Dieu, Paris
  - Hopital St. Antoine, Paris
  - Clinique Saint Hilaire, Rouen
  - Pole de cancerologie prive, Strasbourg
  - CLCC Paul Strauss, Strasbourg
  - Institution Claudius Regaud, Toulouse
  - Polyclinique du Parc, Toulous
- Germany (27):
  - Klinikum St. Marien Amberg, Amberg
  - Hochwaldkrankenhaus, Bad Nauheim
  - Klinikverbund Suedwest - Sindelfingen-Böeblingen Clinical Centre, Böeblingen
  - Klinikum Chemnitz, Chemnitz
  - Universitaetsklinikum Dresden, Dresden
  - Luisenkrankenhaus, Düsseldorf
  - Universitaetsfrauenklinik, Essen
  - Zentrum fur Frauenheilkunde und Geburtshilfe, Frankfurt
  - Medizinisches Versorgungszentrum Osthessen, Fulda
  - Kreiskrankenhaus Hameln, Hamelin
  - Klinikum Stadt Hanau, Hanau
  - Klinikum Hannover Nordstadt, Hanover
  - Universitat Frauenklinik Jena, Jena
  - Onkologische schwerpunktpraxis, Leer
  - Klinikum Lippe Lemgo, Lemgo
  - Asklepios Kliniken Lich GmbH, Lich
  - Universitaetsklinikum Mainz, Mainz
  - St. Vincenz u. Elisabeth Hospital, Mainz
  - Ev Krankenhaus Bethesda, Mönchengladbach
  - RotKreuzKlinikum München GmbH, Munich
  - Universitaetsklinikum Munster, Münster
  - Praxis und Tagesklinik fuer Onkologie und, Recklinghausen
  - Klinikum Rosenheim, Rosenheim
  - Klinikum Schaumburg, Stadhagen
  - Johanniter Krankenhaus, Stendal
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Fachärzte fürlnnere Medizin, Hämatologie, Traunstein
- P.G. Hospital of Thessaloniki "Papageorgiou", Thessaloniki, Greece
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
- Hungary (4):
  - Semmelweis Egyetem Clinic of Radiology, Budapest
  - DEOEC Onkologiai Tanszek, Debrecen
  - Petz Aladar Megyei Oktato, Győr
  - Kaposi Mor oktato korhaz Onkologiai tanszek, Kaposvár
- Ireland (10):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St. James's Hospital, Dublin
  - Adelaide and Meath National Childrens Hospital, Dublin
  - Institute for Cancer Research, Dublin
  - Mater Private Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - University College Hospital Galway, Galway
  - Midwestern Regional Hospital, Limerick
  - Sligo General Hospital, Sligo
- Israel (6):
  - The Lady Davis Carmel Medical Center/Lynn, Haifa
  - Meir Medical Center, Kfar
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Sourasky (Ichilov) Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (11):
  - Humanitas Centro Catanese, Catania
  - (Azienda u.s.I. chieti) - Policinico Ospedaliero, Chieti
  - Ospedale vito fazzi, Lecce
  - Ospedale di Mirano, Mirano
  - IRCCS - Instituto Nazionale per lo Studio e la Cura, Napoli
  - Fondazione Salvatore Maugeri, Pavia
  - Ospedale S. Filippo Neri, Roma
  - Regina Elena Cancer Institute, Rome
  - Ospedale casa sollievo della sofferenza, San Giovanni
  - Universita-istituto Clinica Medica, Sassari
  - Asl n. 5 -Ospedale s. Vincenzo, Taormina
- P. Stradina Clinical University Hospital, Riga, Latvia
- Opcion Oncologia, Monterrey, Mexico
- Peru (2):
  - Hospital Nacional Carlos Alberto Seguin, Arequipa
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
- Cebu Doctors University Hospital, Cebu City, Philippines
- Poland (6):
  - Regional Oncology Center, Bialystok
  - Centrum Onkologii Instytut im. M., Gliwice
  - ZOZ MSWiA z Warminsko-Mazurskim Centrum, Olsztyn
  - Olsztynski Osrodek Onkologiczny "Kopernik", Olsztyn
  - Samodzielny Publiczny Zaklad Opieki, Rybnik
  - Breast Cancer Clinic, Warsaw
- Portugal (2):
  - HUC, Coimbra
  - IPO Francisco Gentil-Porto, Porto
- Romania (3):
  - County Hospital Alba-Iulia, Alba Iulia
  - Institute of Oncology "AI.Trestioreanu", Bucharest
  - Institutul Oncologic "Prof. Dr. I. Chiricuta" Cluj-Napoca, Cluj-Napoca
- Russia (4):
  - State Medical Institution "Republican Clinical Oncology Dispensary Ministry of Health of Republic Tatarstan", Kazan'
  - State Institution "Russian Oncological Research Center n.a. N.N. Blokhin of RAMS", Moscow
  - Federal State Institution "Research Institute of Oncology n.a. N.N. Petrov Rosmedtechnologiy", Saint Petersburg
  - Saint-Petersburg State Medical Institution "City Clinical Oncology Dispensary", Saint Petersburg
- Serbia (2):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinic of Oncology, Clinical Center nis, Niš
- University Clinical Centre, Maribor, Slovenia
- South Africa (3):
  - Department of Oncotherapy National Hospital, Bloemfontein
  - Hopelands Cancer Centre, Durban
  - Johannesburg Hospital, Johannesburg
- South Korea (5):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (38):
  - Hospital Universitario Insular de Gran Canaria, Las Palmas, Canary Islands
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Centro Oncologico de Galicia, A Coruña
  - Fundacion Hospitalaria de Alcorcon, Alcorcón
  - Hospital General de Alicante, Alicante
  - Hospital Perpetuo Socorro, Badajoz
  - Hospital Germans Trias l Pujol, Badalona (Barcelona)
  - Hospital Comarcal de Barbastro, Barbastro
  - Hospital Del Mar, Barcelona
  - Hospital Santa Crue l San Pau, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Consorci Sanitari de Terrassa, Barcelona
  - Althaia Xarxa Assistencial de Manresa, Barcelona
  - Hospital Espiritu Santo, Barcelona
  - Hospital De San Pedro de Alcantara, Cáceres
  - Instituto Oncologico de Guipuzcoa, Donostia / San Sebastian
  - Hospital Gral. De Elche, Elche
  - Hospital de Cabueñes, Oncologia Médica, Gijón
  - Instituto Catalan Oncologia de Girona, Girona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Xera Calde, Lugo
  - Hospital Universitario Gregorio Maranon, Madrid
  - Hospital Ruber International, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Centro Integral de Oncologia "Clara Campal", Madrid
  - Hospital Clinico Virgen de la Victoria, Málaga
  - Hospital Univesitario Carlos Haya, Málaga
  - Hospital Santa Maria Nai Dr. Cabaleiro, Ourense
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital del Parc Tauli, Sabadell
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Torrevieja Salud, UTE, Torrevieja
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital U. Miguel Servet, Zaragoza
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung, Kaohsiung City
  - National Cheng Kung University, Tainan
  - Sun Yat-Sen Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Thailand (3):
  - Chulalongkorn Hospital, Patumwan, Bangkok
  - National Cancer Institute, Bangkok
  - Songklanagarind Hospital, Songkhla
- United Kingdom (7):
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Hematology - Oncology Centre, Bristol
  - Ipswich Hospital, Ipswich
  - Christie Hospital NHS Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Peterborough District Hospital, Peterborough
  - Sunrise Cancer Centre, Truro